CLINICAL TRIAL: NCT00370227
Title: To Assess Safety, Reactogenicity & Immunogenicity of a Booster Dose of Pneumococcal Conjugate Vaccine, Co-admin With GSK Biologicals' MMRV Vaccine in Children (2nd yr of Life) Primed With the Pneumococcal Conjugate Vaccine in Study 105553.
Brief Title: Safety and Immunogenicity Study of a Booster Dose of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107706
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumonia, pneumococcal conjugate vaccine
MeSH Terms: conditions — Streptococcal Infections; Pneumonia | interventions — 10-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 10 valent pneumococcal conjugate (vaccine)

SUMMARY:
This study will evaluate the safety, reactogenicity and immunogenicity of a booster dose of the pneumococcal conjugate vaccine, co-admin with a 1st dose or a 2nd dose of MMRV vaccine at 12-14 or respectively 14-16 months of age in children primed with the pneumococcal conjugate vaccine in study 105553. Antibody persistence will be evaluated at 8-10 months after completion of the 3-dose immunization course in study 105553. The immunogenicity, safety and reactogenicity of the 1st and 2nd dose of MMRV vaccine will also be evaluated when co-admin with the pneumococcal conjugate vaccine between 12-16 months of age.

The study has 3 groups.

* The 1st group will receive the booster dose of pneumococcal conjugate vaccine + 1st dose of MMRV vaccine at 12-14 mo of age and the booster dose of Infanrix hexa™+ 2nd dose of MMRV vaccine at 14-16 mo of age.
* The 2nd group will receive the booster dose of Infanrix hexa™ + 1st dose of MMRV vaccine at 12-14 mo of age and the booster dose of pneumococcal conjugate vaccine + 2nd dose of MMRV vaccine at 14-16 mo of age.
* The 3rd group will receive the booster dose of pneumococcal conjugate vaccine + the booster dose of Infanrix hexa™ at 12-14 mo. Subjects will be offered one dose of Priorix™ and Varilrix™ at 14-16 mo of age, outside the study.

ELIGIBILITY:
Inclusion Criteria:

* a healthy male or female, 12-14 months of age at the time of first vaccination, who received at least one dose of pneumococcal conjugate vaccine during study 105553 and with written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the vaccination, or planned use during the entire study period (active phase and safety follow-up).
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before the first dose of vaccine(s) and ending 42-56 days after the last dose of vaccine(s).
* Administration of any additional pneumococcal vaccine since end of study 105553.
* Previous vaccination against measles, mumps, rubella and/or varicella. History of, or intercurrent measles, mumps, rubella and/or varicella/zoster diseases.
* Known exposure to measles, mumps, rubella and/or varicella/zoster within 30 days prior to study start.
* Immunosuppressive or immunodeficient condition.
* A history of seizures or neurological disease.

Ages: 12 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 390
Dates: Start 2006-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Post vacc: rectal fever >39°C

SECONDARY OUTCOMES:
AEs/ SAEs (42 days/up to 6 mo post last vacc); prior & 42-56 days post vacc: immune response to pneumo & MMRV vaccines antigens.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Finland (7):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Vesikari T, Karvonen A, Lindblad N, Korhonen T, Lommel P, Willems P, Dieussaert I, Schuerman L. Safety and immunogenicity of a booster dose of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine coadministered with measles-mumps-rubella-varicella vaccine in children aged 12 to 16 months. Pediatr Infect Dis J. 2010 Jun;29(6):e47-56. doi: 10.1097/INF.0b013e3181dffabf. PMID 20508478
- [Background] Vesikari T et al. 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine (PHiD-CV) booster co-administered with MMRV vaccine in children aged 12-18 months. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Vesikari T et al. Immunogenicity and safety of a Measles-Mumps-Rubella-Varicella (MMRV) vaccine co-administered with pediatric vaccines in children aged 11-14 months. Abstract presented at the 26th Annual Meeting of the ESPID. Graz, Austria, 13-17 May 2008.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107706 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register